CLINICAL TRIAL: NCT05719350
Title: Effectiveness of Telerehabilitation in Patients With Osteoarthritis. A Randomized Controlled
Brief Title: Telerehabilitation in Patients With Osteoarthritis
Acronym: TABLET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001333
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Tele-rehabilitation exercises for the knee joint to reduce pain
  Interventions: Other: Exercises for Knee
- Control Group (Active Comparator): Exercises in presence for the knee joint to decrease pain
  Interventions: Other: Exercises for Knee

INTERVENTIONS:
Other: Exercises for Knee — Four exercises for strengthening and mobility of the knee joint two in a sitting position and two in a standing position for a total of 20-25 minutes

SUMMARY:
Randomized controlled study on the effectiveness of Telerehabilitation intervention on subjects with knee osteoarthritis. Subjects will be randomized into two groups. The experimental group perform 3 sessions a week for 4 weeks of TR, the control group 3 sessions a week for 4 weeks of conventional rehabilitation c/o IOR rehabilitation gym. Follow-up at 3 months.

Inclusion criteria

1. Subjects must have a diagnosis of rheumatologic disease, osteoarthritis of one or more indications, OARSI criteria.
2. Male or Female, aged > 18 years
3. Participant is willing and able to provide informed consent for participation in the study.
4. Subjects must be able to use an electronic device (pc, tablet, smartphone). Exclusion criteria

1. Participation in another clinical study with any investigational agent within 30 days prior of the study screening.

2. Inability to use an electronic device (pc, tablet, smartphone) 4. Diagnosed with dementia or neurological disease that impairs speech comprehension e Not verbal.

5. Uncontrolled intercurrent illnesses including, without limitation, current infection or active, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illnesses/social situations that would limit compliance with study requirements, illnesses neurological.

6. Children under the age of 18 8. NPRS value <3 7. BMI >25

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of rheumatologic disease, osteoarthritis of one or more articulations, OARSI criteria.
* Male or Female, aged > 18 years
* Participant is willing and able to provide informed consent for participation in the
* study.
* Subjects must be able to use

Exclusion Criteria:

* Participation in another clinical study with any investigational agent within 30 days prior
* of the study screening.
* Inability to use an electronic device (pc, tablet, smartphone)
* Diagnosed with dementia or neurological disease that impairs speech comprehension e Not verbal.
* Uncontrolled intercurrent illnesses including, without limitation, current infection or active, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illnesses/social situations that would limit compliance with study requirements, illnesses neurological.
* hildren under the age of 18
* Numeric Pain Rating Scale(NPRS) value <3
* BMI >25

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
Rating of Pain | one Month
  rating of pain in the knee joint with osteoarthritis measured with the nprs pain scale

SECONDARY OUTCOMES:
Quality of life improvement | one month, three month
  Improved quality of life as measured by the Short Form Health Survey scale
Assessment of knee joint function | one month, three month
  Assessment of knee joint function as measured by the Womac scale

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Benedetti, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Roberto Tedeschi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No